CLINICAL TRIAL: NCT00472875
Title: Do Sulphonylureas Preserve Cortical Function During Hypoglycaemia?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 07/Q0703/18; JDRF grant number 5-2007-478
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2007-05-14 (Estimated); Status verified 2007-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: hypoglycaemia; type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Glibenclamide

SUMMARY:
To see if using medication called sulphonylureas can help improve symptoms which patients rely on to recognise low blood glucose levels ( hypoglycaemia) and also to see if they can reduce the slowing down in brain function which occurs at hypoglycaemia.

DETAILED DESCRIPTION:
Low blood glucose (hypoglycaemia) is the most common and important side effect of insulin treatment for diabetes. Most episodes are "mild" and lead to symptoms that alert the individual to raise their blood sugar level by consuming sugar or starch (carbohydrate). The body also responds to low blood sugars by producing hormones such as adrenaline and cortisol, which help to restore blood sugar levels to normal. As the brain relies on sugar for fuel, it does not function properly if blood sugar levels drop too low, resulting in confusion and in extreme cases reduced conscious levels.

Repeated hypoglycaemia can blunt the protective symptoms and hormonal responses to hypoglycaemia limiting patients' ability to recognise and correct hypoglycaemia, putting them at high risk of even more hypoglycaemia (Heller and Cryer, 1991).

Sulphonylureas are tablets used to treat type 2 diabetes that work by stimulating the pancreas to make more insulin. They do this by closing pores called KATP channels which are found on the surface of many cells and control the rate of firing of cells. In the pancreas, closing them causes cells to fire and release insulin. However, in other tissues such as in the brain, these channels have a protective function and they open up during times of lack of fuel, such as lack of oxygen or sugar, preventing the cells from firing and putting them into a resting mode which reduces their energy requirement(Dunn-Meynell, Rawson and Levin 1998). However, if the brain cells responsible for generating symptoms are put into this resting mode, they may not produce symptoms, which may contribute to hypoglycaemia unawareness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Type 1 diabetes (WHO definition) of at least 5 years duration
* History of impaired awareness of hypoglycaemia (capillary glucose readings < 3.5mmol/l without symptoms on > 3 occasions in the past 3 months (those with intact symptoms will be unlikely to show an improvement and would not really benefit from taking any medication intended just to increase symptoms)

Exclusion Criteria:

* Pregnancy
* Severe systemic illness
* Active malignancy
* Severe complications of diabetes such as severe visual impairment, severe renal impairment, severe symptomatic autonomic neuropathy
* Untreated ischemic heart disease, recent stroke
* Lactose intolerance ( the placebo will contain lactose)
* Very poor diabetes control (HbA1c > 10%) Liver disease ( increase in ALT / AST > 3x ULN)
* Chronic Kidney Disease stage 4 or 5 ( eGFR < 30ml/min)
* Severe untreated thyroid or adrenal insufficiency ( must be treated and on stable doses for at least 6 weeks)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-05

PRIMARY OUTCOMES:
Glucose threshold for development of symptoms and cognitive impairment due to hypoglycaemia | 1 year

SECONDARY OUTCOMES:
Improvement in counter regulatory hormone response to hypoglycaemia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pratik Choudhary, MBBS MRCP, Principal Investigator — King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom